CLINICAL TRIAL: NCT05440097
Title: Change Asthma Clinical Practice Through Guideline Education and Implementation For All Patients With Asthma: an Evaluation of an Asthma Quality Improvement Program
Brief Title: CARE FOR ALL：an Evaluation of an Asthma QIP
Acronym: CARE FOR ALL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D589BC00027
Record Dates: First submitted 2022-06-02; First posted 2022-06-30 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm (Other): GINA guideline education and implementation
  Interventions: Other: QIP intervention

INTERVENTIONS:
Other: QIP intervention — The QIP includes pulmonologist-targeted guideline education and guideline implementation.
  Guideline education includes the initial comprehensive training and reinforcement learning. The initial comprehensive education will be delivered at each participating hospital by a dedicated national asthma expert team, immediately after last patient enrolled at each site. The PI of respiratory departments from participating hospitals are responsible for arranging the delivery of hospital-level reinforcement learnings and ensuring the quality and success of hospital-level guideline implementation.
  The pulmonologists' guideline adherence and performance at participating hospitals will be regularly assessed during the study period.

SUMMARY:
This is an evaluation on an asthma Quality Improvement Program (QIP, including GINA guideline education/training and implementation) to understand the change of physician behaviours, which leads to the change of patient outcomes. Primary endpoint is "Change from baseline in the proportion of participants with an ICS-based maintenance and/or reliever treatment at week 48 ".

A total of around 30 eligible Tier 3 and Tier 2 hospitals will be selected across China. Approximately 1500 eligible asthmatic patients fulfilling the following inclusion and exclusion criteria will be enrolled consecutively from participating hospitals,.

The QIP (including GINA guideline education/training and implementation) will be delivered at the hospital level, targeting all pulmonologists and specialist nurses at participating hospitals, including initial comprehensive education, reinforcement learning, and performance assessment and feedback of pulmonologists' guideline implementation, along with multiple online and offline approaches serving as reminders and supportive tools to ensure consistent education and to facilitate the asthma management in routine clinical practice in accordance with GINA recommendation.

After the initiation of the intervention program participating patients will return to the study hospital every 12 weeks for on-site follow-up visits (V1 to V5), in accordance with guideline recommendations. Meanwhile, investigators are mandatory requested to join in reinforce education at regular time. Guideline implementation performance will be assessed against with multi-approach indicators for each participant's offline or online visit.

The objective of the CARE FOR ALL study is to bridge the gap that exists between the recommendations from GINA 2021 and current clinical practice by demonstrating the benefits of an asthma quality improvement program (QIP), i.e. a standardized pulmonologist-targeted GINA guideline education and practice implementation.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 14 years of age or older at the time of signing the informed consent.
2. Physician-confirmed asthma diagnosis with documented evidence of variable expiratory airflow limitation (e.g. from bronchodilator reversibility testing or other test)
3. Participating patients and/or their legally authorised representative must provide signed and dated written informed consent form prior to any study specific procedures.

Exclusion Criteria:

1. Previous diagnosis of chronic obstructive pulmonary disease (COPD) or other clinically relevant chronic respiratory disease other than asthma
2. Any significant disease or disorder (e.g. cardiovascular, pulmonary other than asthma, gastrointestinal, hepatic, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment) which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or may influence the results of the study, or the patient's ability to participate in the study
3. Disease or condition other than asthma that requires treatment with systemic or oral steroids
4. Participation in another clinical study with an Investigational Product administered in the last 3 months prior to Visit 1.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- China (29):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Changzhi
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Foshan
  - Research Site, Guangzhou
  - Research Site, Handan
  - Research Site, Harbin
  - Research Site, Hebi
  - Research Site, Hefei
  - Research Site, Huai'an
  - Research Site, Jinan
  - Research Site, Jinhua
  - Research Site, Kunming
  - Research Site, Kunshan
  - Research Site, Nanchang
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shiyan
  - Research Site, Taizhou
  - Research Site, Tianjin
  - Research Site, Wuhu
  - Research Site, Wuyishan
  - Research Site, Xi'an
  - Research Site, Yantai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Huang K, Wang W, Wang Y, Li Y, Feng X, Shen H, Wang C. Evaluation of a Global Initiative for Asthma Education and Implementation Program to Improve Asthma Care Quality (CARE4ALL): Protocol for a Multicenter, Single-Arm Study. JMIR Res Protoc. 2025 Jan 8;14:e65197. doi: 10.2196/65197. PMID 39778197
- See also: D589BC00027_Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D589BC00027&attachmentIdentifier=0da33007-2c88-4b43-970c-cef4bea8e3c8&fileName=D589BC00027_CSP_Redacted.pdf&versionIdentifier=
- See also: D589BC00027_Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D589BC00027&attachmentIdentifier=7ea59f6c-faf6-4bb2-b01a-768d5ce5397f&fileName=D589BC00027_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: D589BC00027_Redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D589BC00027&attachmentIdentifier=56f49eae-1ef6-491a-a3bc-41c70c251f00&fileName=D589BC00027_SAP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-arm study assessed a hospital-level Quality Improvement Program (QIP) in 31 Chinese hospitals (29 Jul 2022 - 03 Sep 2024). The QIP was a standardized GINA 2021 guideline education intervention delivered to 282 engaged pulmonologists. Participant Population (Outcome Assessors): Consecutive asthma patients from these hospitals were screened; 1,536 were screened and 1,500 were enrolled to be managed by the trained pulmonologists.
Pre-assignment Details: For Pulmonologists: All participating pulmonologists from the 31 hospitals received the QIP intervention. There was no control group of pulmonologists .Baseline data were not collected for Pulmonologists. For Patients: All enrolled patients were managed by pulmonologists who had received the QIP. Patients were not randomized to different treatment strategies; the study aimed to observe the change in their outcomes before and after their physicians received the QIP.
Groups:
- Total: Total of all participants
Period: Overall Study
Arm/Group | Total
Started | 1500
Full Analysis Set (All enrolled participants with at least one non-missing post-intervention GINA guideline treatment assessment.) | 1362
Completed | 1271
Not Completed | 229
Not completed — Withdrawal by Subject | 154
Not completed — Death | 2
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 56
Not completed — Include "enrolled by mistake" and "withdrawed by mistake". | 15

BASELINE CHARACTERISTICS:
Population: 1,362 patients were included in the FAS. All analyses were conducted based on FAS.
Arm/Group | Total
Number analyzed (Participants) | 1362
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (14.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 800
  Male | 562
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1362
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Proportion of Patients With an ICS-based Maintenance and/or Reliever Treatment
Description: Change from baseline in the proportion of patients with an ICS-based maintenance and/or reliever treatment at week 48 was performed using mixed effect logistic regression model.
Time Frame: Baseline to week 48
Population: All successfully enrolled participating patients were followed up for up to 48 weeks and returned to recruiting hospital for study visits every 12 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Full Analysis Set: All enrolled participants with at least one non-missing post-intervention GINA treatment assessment were enrolled into FAS.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 1362
Participants
  Baseline | 571
  Week 48: number analyzed (Participants) | 1314
  Week 48 | 723
Statistical Analysis 1: Comparison: Full Analysis Set; Test type: Other; p < .0001, Mixed Models Analysis; The primary analysis used mixed effect logistic regression model, taking the timepoint as the fixed effect, hospital and patient as random effects; Difference in percentage = 12.79, 95% CI 2-sided [9.079 to 13.431]

2. Secondary Outcome: Secondary Endpoint 1- Change From Baseline in the Proportion of Participants With Well-controlled Asthma (ACQ-5 ≤ 0.75) at Week 48
Description: The Asthma Control Questionnaire-5 (ACQ-5) is a shortened version of the full 7-item ACQ (Juniper et al 1999) that assesses asthma symptoms (night-time awakening, symptoms on awakening, activity limitation, shortness of breath, and wheezing). Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-5 score is the mean of the responses. Mean scores of ≤0.75 indicate well controlled asthma, 0.75-1.5 indicate partly controlled asthma, and ≥1.5 indicates not well controlled asthma.
Time Frame: Baseline to Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 1362
Participants
  Baseline: number analyzed (Participants) | 1357
  Baseline | 354
  Week 48: number analyzed (Participants) | 1132
  Week 48 | 641
Statistical Analysis 1: Comparison: Full Analysis Set; Test type: Superiority; Normal approximation; Difference in percentage = 30.5, 95% CI 2-sided [26.82 to 34.25]

3. Secondary Outcome: Secondary Endpoint 2- Change From Baseline in the Proportion of Patients on the Treatment of ICS-formoterol as Reliever at Week 12, 24, 36 and 48
Time Frame: Baseline, week 12, 24, 36 and 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 1362
Participants
  Baseline: number analyzed (Participants) | 491
  Baseline | 2
  Week 12: number analyzed (Participants) | 581
  Week 12 | 15
  Week 24: number analyzed (Participants) | 485
  Week 24 | 12
  Week 36: number analyzed (Participants) | 508
  Week 36 | 64
  Week 48: number analyzed (Participants) | 624
  Week 48 | 84
Statistical Analysis 1: Comparison: Full Analysis Set; Test type: Superiority; Normal approximation; Difference in percentage = 2.2, 95% CI 2-sided [0.77 to 3.58] — Change from baseline in proportion at week 12
Statistical Analysis 2: Comparison: Full Analysis Set; Test type: Superiority; Normal approximation; Difference in percentage = 2.1, 95% CI 2-sided [0.57 to 3.56] — Change from baseline in proportion at week 24
Statistical Analysis 3: Comparison: Full Analysis Set; Test type: Superiority; Normal approximation; Difference in percentage = 12.2, 95% CI [9.25 to 15.13] — Change from baseline in proportion at week 36
Statistical Analysis 4: Comparison: Full Analysis Set; Test type: Superiority; Normal approximation; Difference in percentage = 13.1, 95% CI [10.32 to 15.79] — Change from baseline in proportion at week 48

4. Secondary Outcome: Secondary Endpoint 3- Change From Baseline in ACQ-5 Average Score at Week 12, 24, 36 and 48
Description: The Asthma Control Questionnaire-5 (ACQ-5) is a shortened version of the full 7-item ACQ (Juniper et al 1999) that assesses asthma symptoms (night-time awakening, symptoms on awakening, activity limitation, shortness of breath, and wheezing). Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-5 score is the mean of the responses.
Time Frame: Baseline, week 12, 24, 36 and 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 1362
Scores on a scale
  Week 12: number analyzed (Participants) | 1138
  Week 12 | -0.59 (1.132)
  Week 24: number analyzed (Participants) | 1142
  Week 24 | -0.65 (1.168)
  Week 36: number analyzed (Participants) | 1117
  Week 36 | -0.61 (1.142)
  Week 48: number analyzed (Participants) | 1130
  Week 48 | -0.71 (1.132)

5. Secondary Outcome: Secondary Endpoint 4- Change From Baseline in the Proportion of Participants With an ICS-based Maintenance and/or Reliever Treatment at Week 12, 24 and 36
Time Frame: Baseline, week 12, 24 and 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 1362
Participants
  Baseline | 571
  Week 12: number analyzed (Participants) | 1232
  Week 12 | 677
  Week 24: number analyzed (Participants) | 1245
  Week 24 | 577
  Week 36: number analyzed (Participants) | 1218
  Week 36 | 590
Statistical Analysis 1: Comparison: Full Analysis Set; Test type: Superiority; Normal approximation; Difference in percentage = 13.0, 95% CI 2-sided [9.21 to 16.85] — Change from baseline in the Proportion at week 12
Statistical Analysis 2: Comparison: Full Analysis Set; Test type: Superiority; Normal approximation; Difference in percentage = 4.4, 95% CI 2-sided [0.61 to 8.23] — Change from baseline in the proportion at week 24
Statistical Analysis 3: Comparison: Full Analysis Set; Test type: Superiority; Normal approximation; Difference in percentage = 6.5, 95% CI 2-sided [2.68 to 10.36] — Change from baseline in the proportion at week 36

ADVERSE EVENTS:
Description: Adverse Event were not collected as part of this study.
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The Institution shall own all rights and title in and to the StudyDocumentation. Inacknowledgment of the contribution made by AstraZeneca to the Study, the Institution shall disclose all or any portion of the Study Documentation to AstraZeneca on request, and shall permit AstraZeneca to use the disclosed Study Documentation for any purpose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT05440097/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT05440097/SAP_001.pdf